CLINICAL TRIAL: NCT00132158
Title: A Dose Finding Study (Phase I) of the Combination of ZD1839 (Iressa®) and an Oral Formulation of Irinotecan (Camptosar™) in Children With Refractory Solid Tumors
Brief Title: ZD1839 and Oral Irinotecan in Treating Young Patients With Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POCPZD; IRUSIRES0181 (Other: AstraZeneca)
Record Dates: First submitted 2005-08-17; First posted 2005-08-19 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: Glioblastoma; Rhabdomyosarcomas; Neuroblastoma; Osteosarcoma
MeSH Terms: conditions — Glioblastoma; Rhabdomyosarcoma; Neuroblastoma; Osteosarcoma | interventions — Irinotecan; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Drug: Irinotecan (Camptosar), Gefitinib (Iressa)

INTERVENTIONS:
Drug: Irinotecan (Camptosar), Gefitinib (Iressa) — See Detailed Description for treatment plan.

SUMMARY:
The purpose of this Phase I study is to find the largest dose of the drug irinotecan, in combination with ZD1839, that can be given safely to children and to learn the good and bad effects. Studies performed in the laboratory have shown that ZD1839 helps make available the orally administered irinotecan. In this study the intravenous (given into the vein) formula of irinotecan will be given orally on days 1-5 and days 8-12. The dose of ZD1839 will be a fixed dose and will be administered orally on days 1-12. Each course of treatment will consist of 21 days. The administration of irinotecan on day 12 of course 1 and day 2 of course 2 will be an intravenous administration. All other doses and subsequent courses will consist of an orally administered dose.

DETAILED DESCRIPTION:
This is a phase I study to estimate the maximum tolerated dose and the dose limiting toxicities of the intravenous formulation of irinotecan given orally in combination with a fixed dose of oral gefitinib. This trial will use the EWOC method, which is an adaptive dose escalation scheme. The method is fully adaptive and makes use of all the information available at the time of each dose assignment, and directly addresses the ethical need to control the probability of overdosing. It is designed to approach the maximum tolerated dose (MTD) as fast as possible.

In this study the intravenous formulation of irinotecan will be given orally on days 1-5 and days 8-12 (dose level begins at 5 mg/m2 ). One patient will be treated at each dose level of irinotecan until moderate toxicity is observed. At the level where moderate toxicity is observed, the cohort size will be increased to 2 patients. Dosages will then be increased until the development of DLT as guided by the EWOC model. The estimated MTD will be continually reassessed using all data from preceding patients. The toxicity data of all patients enrolled in the trial are used to update the dose-toxicity relationship and to guide the next escalation/de-escalation. The calculation will be carried out with EWOC software. Patients will be enrolled and the dose assigned is determined based on previous participants' toxicity. The dose of ZD1839 will be a fixed dose and will be administered orally on days 1-12 - [150 mg/m2 (maximum 250 mg)] Each course of treatment will consist of 21 days. The administration of irinotecan on day 12 of course 1 and day 2 of course 2 will be an intravenous administration. All other doses and subsequent courses will consist of an orally administered dose.

Secondary Objectives Include:

* To describe dose-limiting toxicities (DLTs) of the combination of oral irinotecan and ZD1839 and to define their duration and reversibility.
* To investigate the pharmacokinetics of oral irinotecan and ZD1839 when given in combination in children with recurrent malignant solid tumors.
* To describe the relationship between pharmacokinetic parameters and toxicity.
* To describe any antitumor effects within the confines of a phase I study.
* To examine tumor expression of ErbB1 and/or ABCG2 with respect to pharmacokinetics and response.
* To examine the pharmacogenetic determinants of ZD1839 and irinotecan pharmacokinetics and pharmacodynamics.

ELIGIBILITY:
Inclusion Criteria:

* Patient's age is less than or equal to 21 years at the time of study entry.
* Patient has a histologically or pathologically confirmed diagnosis of a recurrent solid tumor that did not respond to standard treatment or one for which there is no known therapy.
* Patient has adequate performance status, along with adequate function of the liver, kidney and bone marrow.
* Must have recovered from chemotherapy
* No active GVHD nor treatment for GVHD

Exclusion Criteria:

* Patient is receiving other cytotoxic or investigational drug or has evidence of another active illness
* Active diarrhea
* Active intercurrent serious or uncontrolled illness
* Pregnant or lactating
* Concomitant use of medications that may interact with study drugs
* Active infection
* Known history of life-threatening allergy or hypersensitivity to camptothecin Active interstitial lung disease

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2005-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To estimate the maximum tolerated dose (MTD) of the intravenous formulation of irinotecan given orally in combination with a fixed dose of oral gefitinib. | Within the first 30 days of completion of first cycle of chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M McGregor, MD, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org